CLINICAL TRIAL: NCT04725331
Title: A Phase I/IIa Study of Intra-tumoral BT-001 (TG6030) Administered Alone and in Combination With Pembrolizumab in Patients With Cutaneous or, Subcutaneous Lesions or Easily Injectable Lymph Nodes of Metastatic/Advanced Solid Tumors.
Brief Title: A Clinical Trial Assessing BT-001 Alone and in Combination With Pembrolizumab in Metastatic or Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision following completion of Phase I part not driven by safety reason
Sponsor: Transgene (Industry)
Collaborators: BioInvent International AB (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BT-001.01; 2020-000505-80 (EudraCT Number); MK3475-E37 (Other: Merck Sharp & Dohme LLC); KEYNOTE-E37 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2021-01-25; First posted 2021-01-26 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Cancer; Soft Tissue Sarcoma; Merkel Cell Carcinoma; Melanoma; Triple Negative Breast Cancer; Non Small Cell Lung Cancer
Keywords: Superficial tumors; Metastatic cancer; Intratumoral; Safety; Oncolytic virus; Vaccinia virus; Solid tumors; Melanoma; Merkel; Sarcoma; TNBC; NSCLC; Pembrolizumab; BT-001; TG6030; Phase 1
MeSH Terms: conditions — Neoplasm Metastasis; Sarcoma; Carcinoma, Merkel Cell; Melanoma; Triple Negative Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Vaccinia | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase I, Part A - Dose escalation and safety of BT-001 alone (Experimental): Dose escalation with repeated administrations of BT-001 directly into tumor as a single agent, in patients with metastatic or advanced solid tumors.
  Interventions: Biological: BT-001
- Phase I, Part B - Safety of BT-001 in combination with pembrolizumab (Experimental): Repeated administrations of BT-001 directly into tumor in combination with infusions of pembrolizumab in patients with metastatic or advanced soft tissue sarcoma (STS), Merkel cell carcinoma (MCC), melanoma, triple negative breast cancer (TNBC) or non-small cell lung cancer (NSCLC)..
  Interventions: Biological: BT-001; Drug: Pembrolizumab [KEYTRUDA®]
- Phase IIa - Expansion cohorts of BT-001 in combination with pembrolizumab (Experimental): Repeated administrations of BT-001 directly into tumor in combination with infusions of pembrolizumab in several cohorts of patients with defined metastatic or advanced solid tumor conditions: soft tissue sarcoma, Merkel cell carcinoma, melanoma, triple negative breast cancer, non-small cell lung cancer.
  Interventions: Biological: BT-001; Drug: Pembrolizumab [KEYTRUDA®]

INTERVENTIONS:
Biological: BT-001 — Oncolytic Vaccinia virus containing genes encoding the 4-E03 human recombinant anti-hCTLA4 antibody and human GM-CSF administered at different dose [Phase I, Part A]; one dose lower and at Recommended Dose for Part B [Phase I, Part B] by intra-tumoral (IT) route.
Drug: Pembrolizumab [KEYTRUDA®] — Programmed death receptor (PD-1) blocking antibody administered at 200mg by intravenous (IV) infusions every 3 weeks.
  Other Names: KEYTRUDA®
  Arms: Phase I, Part B - Safety of BT-001 in combination with pembrolizumab; Phase IIa - Expansion cohorts of BT-001 in combination with pembrolizumab

SUMMARY:
This is a Phase I/IIa, multicenter, open-label, consecutive cohorts, dose-escalation study of BT-001 with repeated IT administrations alone and in combination with IV infusions of pembrolizumab.

DETAILED DESCRIPTION:
This study will include 3 parts:

* Phase I, Part A: Repeated intra-tumoral (IT) administrations of BT-001 as a single agent, in patients with metastatic/advanced solid tumors; dose-escalation will be employed.
* Phase I, Part B: Repeated IT administrations of BT-001 in combination with intravenous (IV) infusions of pembrolizumab in patients with metastatic/advanced soft tissue sarcoma (STS), Merkel cell carcinoma (MCC), melanoma, triple negative breast cancer (TNBC) or non-small cell lung cancer (NSCLC)..
* Phase IIa: Repeated IT administrations of BT-001 in combination with IV infusions of pembrolizumab in several cohorts of patients with defined metastatic or advanced solid tumor conditions.

ELIGIBILITY:
Inclusion Criteria:

* Have at least 1 injectable measurable cutaneous, subcutaneous or nodal lesion (direct injection or through the use of ultrasound guidance) not exceeding 50mm in longest diameter and whenever possible 1 distant non-injected measurable lesion.
* Provision of a fresh tumor sample of the lesion that will be injected first and, whenever possible, from another lesion that is planned to be injected, at baseline and be willing to supply new tumor samples from a biopsy during treatment.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1.
* Have adequate hematological, hepatic and renal functions.
* Have histologically confirmed, advanced/metastatic sarcoma (soft tissue and bone), Merkel cell carcinoma, melanoma, triple negative breast cancer or non-small cell lung cancer, with cutaneous or, palpable subcutaneous lesions or easily injectable lymph nodes.
* Have failed and/or are intolerant to standard therapeutic options.

Exclusion Criteria:

* Have had major surgery within 4 weeks of first study drug administration.
* Have received prior treatment with a vaccinia oncolytic virus.
* Have received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to the start of treatment.
* Have received prior radiotherapy within 2 weeks of start of study treatment or have had a history of radiation pneumonitis
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 28 days prior the first dose of study drugs
* Have a known additional malignancy that is progressing or has required active treatment within the past 3 years.
* Have an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs).
* Have a history of (non-infectious) pneumonitis / interstitial lung disease that required steroids or has current pneumonitis / interstitial lung disease
* Have an active infection requiring systemic therapy
* Have a known history of HIV infection
* Is taking an anticoagulant medication that cannot be interrupted prior to IT injections
* Have had an allogenic tissue/solid organ transplant or allogenic stem cell or bone marrow transplantation
* History of severe exfoliative skin conditions (e.g., eczema or atopic dermatitis) requiring systemic therapy for more than 4 weeks within 2 years prior to BT-001 initiation.
* Have received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137), and was discontinued from that treatment due to a Grade 3 or higher immune-related Adverse Event (irAE).
* Have known active CNS metastases and/or carcinomatous meningitis.
* Have a known history of Hepatitis B (defined as HBsAg reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection.n.
* Woman of childbearing potential who has a positive serum pregnancy test (within 72 hours) prior to the start of treatment.
* Have received or receiving any live or live-attenuated vaccine within 30 days prior to the first dose of study intervention..
* History of myocarditis or congestive heart failure, unstable angina, uncontrolled infection, or myocardial infarction 6 months prior to clinical trial entry.
* Interstitial lung disease that is symptomatic and may interfere with the detection or management of suspected drug-related pulmonary toxicity
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment
* Have severe hypersensitivity to the active substance or, to any of the excipients of (≥Grade 3) to pembrolizumab. and/or any of its excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2025-10-22 (Actual); Study Completion 2025-10-22 (Actual)

PRIMARY OUTCOMES:
Phase I: Safety and tolerability (Adverse Event reported per NCI-CTCAE v5.0) | Up to 5 years
  Incidence of Adverse Event reported per NCI-CTCAE v5.0, Dose limiting toxicity and Serious Adverse Events.
Phase I, Part A: Recommended dose for Part B (RDPB) definition | Week 10-12
  RDPB based on the safety data collected during the dose escalation phase (Phase I, Part A).
Phase IIa (except Soft Tissue Sarcoma cohort): Immune Overall Response Rate (iORR) by iRECIST | Up to 2 years
  Percentage of patients whose best overall response is either a Complete Response or a Partial Response according to immune Response Evaluation Criteria In Solid Tumors (iRECIST) criteria over the the total number of evaluable patients. for injected and non-injected lesion(s)
Phase IIa (Soft Tissue Sarcoma cohort): Immune Disease Control Rate (iDCR) at 6 months by iRECIST | Up to 6 months
  Percentage of patients whose best overall response is either a Complete Response, a Partial Response or Stable Disease according to immune Response Evaluation Criteria In Solid Tumors (iRECIST) criteria over the the total number of evaluable patients.

SECONDARY OUTCOMES:
Phase IIa: Safety and tolerability (Adverse Event reported per NCI-CTCAE v5.0) | Up to 5 years
  Incidence of Adverse Event reported per NCI-CTCAE v5.0, Dose limiting toxicity and Serious Adverse Events.
Disease Control Rate (DCR) and immune DCR by RECIST version 1.1 and iRECIST | 4 months or 6 months
  Percentage of patients whose best overall response is either a Complete Response, a Partial Response or Stable Disease according to Response Evaluation Criteria In Solid Tumors version 1.1 (RECIST 1.1) criteria or immune RECIST over the total number of evaluable patients.
Progression Free Survival (PFS) and immune PFS duration by RECIST version 1.1 and iRECIST | Up to 2 years
  Time from the first BT-001 administration to the date of first documented tumor progression according to Response Evaluation Criteria In Solid Tumors version 1.1 (RECIST 1.1) criteria or immune RECIST or death due to any cause, whichever occurs first over evaluable patients
Duration of overall Response (DoR) and immune DOR by RECIST version 1.1 and iRECIST | Up to 2 years
  Time from the date of first documented response (CR or PR) to the date of first documented disease progression according to Response Evaluation Criteria In Solid Tumors version 1.1 (RECIST 1.1) criteria or immune RECIST or the date of death due to underlying cancer over the number of patients whose Best Overall Response is Complete Response or Partial Response.
Overall Survival (OS) duration | Up to 2 years
  Time from first BT-001 administration to the date of death due to any cause over evalauable patients.

CONTACTS AND LOCATIONS:
Locations (5):
- Clinique Universitaire Saint-Luc, Brussels, Belgium
- France (4):
  - Institut Bergonié, Bordeaux
  - Centre Léon Bérard, Lyon
  - Hôpital Saint-Louis AP-HP, Paris
  - Institut Gustave Roussy, Villejuif